CLINICAL TRIAL: NCT03366116
Title: Phase I Trial of 5-aza-4'-Thio-2'-Deoxycytidine (Aza-TdC) in Patients With Advanced Solid Tumors
Brief Title: 5-aza-4'-Thio-2'-Deoxycytidine (Aza-TdC) in People With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 180014; 18-C-0014
Record Dates: First submitted 2017-12-07; First posted 2017-12-08 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01-22

CONDITIONS: Neoplasms; Solid Tumors
Keywords: Pharmacodynamics; DNA Methylation; Pharmacokinetics; Nucleoside Analog; Epigenetics
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Aza-TdCyd will be administered orally once a day for 5 days of each week for 2 weeks, with one week off, in 21-day cycles
  Interventions: Drug: aza-TdC

INTERVENTIONS:
Drug: aza-TdC — Methylation-mediated silencing of genes is an epigenetic mechanism implicated in carcinogenesis; agents that inhibit this mechanism are of clinical interest because of their potential to re-activate silenced tumor suppressor genes. The nucleoside analog 5-aza-4'-thio-2'- deoxycytidine (Aza-TdC) is incorporated into DNA, where it engages the active site of DNA methyltransferase I (DNMT1), a maintenance methyltransferase that contributes to hypermethylation and silencing of tumor suppressor genes. Aza-TdC offers an improvement over traditional DNMT inhibitors via higher incorporation into DNA and lower cytotoxicity; Aza-TdC has greater antitumor activity than another recently developed DNMT1 inhibitor, TdCyd, in some solid tumor xenograft models. Treatment with Aza-TdC is anticipated to yield inhibition of tumor growth due to DNMT1 depletion at oral doses that are well tolerated in extended dosing schedules.

SUMMARY:
Background:

Blood, tissue, and tumor cells contain genes. Genes are made up of DNA. DNA is the "instruction book" for each cell. In some people with cancer, the genes that might have slowed the growth of their tumor were "turned off." Researchers want to see if a new drug can turn the genes back on and slow the tumor growth. The drug is called Aza-TdC.

Objective:

To test the safety of Aza-TdC, and to find out the dose of this drug that can be safely given to humans.

Eligibility:

People ages 18 and older who have advanced cancer that has gotten worse after standard treatment, or for which no effective therapy exists

Design:

Participants will be screened with:

Medical history

Blood and urine tests

Scans to measure their tumors

Test to measure the electrical activity of the heart

Participants will take the study drug by mouth. The drug is given in cycles. Each cycle is 21 days (3 weeks) long.

Week 1 and week 2: participants will take the study drug once a day for 5 days. Then they will have 2 days without the drug. Week 3: no study drug is taken. This completes one cycle of treatment.

For cycle 1, participants will repeat the screening tests several times. For all other cycles, participants will have blood tests and pregnancy tests. They will have scans of their tumor every 6 weeks.

The cycle will be repeated as long as the participant tolerates the drug and the cancer is either stable or gets better.

Sponsoring Institute: National Cancer Institute

DETAILED DESCRIPTION:
Background:

Methylation-mediated silencing of genes is an epigenetic mechanism implicated in carcinogenesis; agents that inhibit this mechanism are of clinical interest because of their potential to re-activate silenced tumor suppressor genes. Two DNA hypomethylating nucleosides, 5-azacytidine (azacytidine) and 5-aza-2'-deoxycytidine (decitabine) have been approved by the FDA for the treatment of patients with myelodysplastic syndromes and certain leukemias.

The nucleoside analog 5-aza-4 -thio-2 -deoxycytidine (Aza-TdC) is incorporated into DNA, where it engages the active site of DNA methyltransferase I (DNMT1), a maintenance methyltransferase that contributes to the hypermethylation and silencing of tumor suppressor genes. DNMT1 can become trapped in a covalent complex with DNA, thus depleting free enzyme and inhibiting the normal maintenance methylation of CpG sites, resulting in re-activation of tumor suppressor genes.

Data suggest a correlation between Aza-TdC activity in solid tumor xenograft models and decreased levels of DNMT1.

Aza-TdC offers an improvement over traditional DNA methyltransferase inhibitors by virtue of a higher incorporation rate into DNA at lower levels of cytotoxicity; Aza-TdC has greater antitumor activity than another recently developed DNMT1 inhibitor, TdCyd, in some solid tumor xenograft models. Treatment with Aza-TdC is anticipated to result in the inhibition of tumor growth due to DNMT1 depletion at oral doses that are well tolerated in extended dosing schedules.

Primary Objective:

To establish the safety, tolerability, and MTD of oral Aza-TdC administered daily for 5 days a week for 2 weeks, with one week off, q 21-day cycles, to patients with refractory solid tumors

Secondary Objectives:

To determine the pharmacokinetics of oral Aza-TdC

To document preliminary evidence of Aza-TdC activity

To determine effect of study treatment on re-expression of select genes silenced by methylation in circulating tumor cells

To determine the effects of Aza-TdC on DNA damage response (DDR) signaling and on genome-wide DNA methylation in tumor biopsy tissue

Exploratory Objective:

To determine the effects of Aza-TdC on global RNA expression and on levels of DNMT1, DNMT3a, DNMT3b, and other select proteins in tumor biopsy tissue

To examine genomic alterations in circulating tumor DNA (ctDNA) that may be associated with Aza-TdC response or resistance

Eligibility:

Patients >= 18 years of age must have histologically documented solid tumors whose disease has progressed on standard therapy or for which there is no available standard therapy

Study Design:

Aza-TdC will be administered orally once a day for 5 days of each week for 2 weeks, with one week off, in 21-day cycles.

The trial will follow an accelerated titration design, changing to a traditional 3+3 dose escalation design (3-6 patients per cohort) once specified toxicity criteria are met. Intrapatient dose escalation will be allowed.

Blood samples will be obtained for pharmacokinetic analysis and to isolate circulating tumor cells to assess re-expression of genes silenced by methylation.

Up to 21 patients will be accrued to a PD expansion cohort at the MTD to further assess pharmacodynamic endpoints in tumor and blood.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically documented solid tumors whose disease has progressed on standard therapy or for which there is no available standard therapy.
* Age >=18 years of age.
* ECOG performance status <= 2.
* Patients must have normal organ and marrow function as defined below:

  * absolute neutrophil count >= 1,500/mcL
  * platelets >=100,000/mcL
  * total bilirubin <=1.5 X institutional upper limit of normal (<=3 x upper limit of normal in the presence of documented Gilbert s syndrome)
  * AST(SGOT)/ALT(SGPT) <=3 X institutional upper limit of normal

OR

* AST(SGOT)/ALT(SGPT) <=5 X institutional upper limit of normal for patients with liver metastases
* creatinine <=1.5X institutional upper limit of normal

OR

* creatinine clearance >=60 mL/min/1.73 m^2 for patients with creatinine levels above 1.5X institutional normal

  * Because nucleoside analogs are known to be teratogenic, women of child-bearing potential and men must agree to use two forms of contraception (hormonal or barrier method of birth control; abstinence; sterilization) prior to study entry, for the duration of study participation, and for 3 months after completing study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use two forms of contraception prior to the study, for the duration of study participation, and for 3 months after completion of administration of Aza-TdC.
  * Patients must have completed any chemotherapy or biologic therapy >= 4 weeks or 5 half-lives (whichever is shorter) (6 weeks for nitrosoureas or mitomycin C) prior to entering the study. Patients must be >= 2 weeks since any prior palliative radiation or cyberknife therapy. Patients must have recovered to grade 1 from prior toxicity or adverse events. Patients on study may be eligible for palliative radiotherapy to non-targeted lesions after 2 cycles of therapy at the PI's discretion. Patients with bone metastases or hypercalcemia on intravenous bisphosphonate treatment prior to study entry may continue this treatment.
  * Ability to understand and the willingness to sign a written informed consent document.
  * Willingness to provide blood and urine samples for research purposes.
  * Ability to swallow pills/capsules.
  * Left ventricular ejection fraction greater than 45% or the institutional lower limit of normal by either ECHO or MUGA at entry.
  * For patients enrolled on the expansion cohort, patients must have tumor amenable to biopsy (excisional or incision biopsies of skin or H & N lesions under visualization) and willingness to undergo tumor biopsies.

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agents.
* Pregnant women and women who are breastfeeding are excluded from this study.
* Patients with clinically significant illnesses which would compromise participation in the study, including, but not limited to active or uncontrolled infection, immune deficiencies, known HIV infection requiring protease inhibitor therapy, known Hepatitis B, known Hepatitis C, uncontrolled diabetes, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with known primary central nervous system (CNS) malignancy or symptomatic CNS metastases are excluded, with the following exceptions:

  * Patients with asymptomatic untreated CNS disease may be enrolled, provided all of the following criteria are met:

    * Evaluable or measurable disease outside the CNS
    * No metastases to brain stem, midbrain, pons, medulla, or cerebellum
    * No history of intracranial hemorrhage or spinal cord hemorrhage
    * No ongoing requirement for dexamethasone for CNS disease; patients on a stable dose of anticonvulsants are permitted.
    * No neurosurgical resection or brain biopsy within 28 days prior to Cycle 1, Day 1
  * Patients with treated CNS metastases may be enrolled, provided all the criteria listed above are met as well as the following:

    * No stereotactic radiation or whole-brain radiation within 14 days prior to Cycle 1, Day 1
    * Screening CNS radiographic study 2 weeks from completion of radiotherapy and >=1 week from discontinuation of corticosteroids. The presence of new CNS mets will not exclude the patient but provide a baseline. If the irradiated lesion showed increased edema or growth, patient may be enrolled if asymptomatic but a repeat MRI should be done within the next 2-4 weeks for follow up.
* Malabsorption syndrome or other conditions that would interfere with intestinal absorption.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2018-11-05 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
To determine the safety, tolerability, and MTD of oral aza-TdCyd administered daily for 5 days a week for 2 weeks, with one week off, in 21-day cycles | Cycle 1 and Cycle 2
  To determine the safety, tolerability, and MTD of oral aza-TdC administered daily for 5 days a week for 2 weeks, with one week off, in 21-day cycles

SECONDARY OUTCOMES:
To determine the pharmacokinetics of oral aza-TdCyd | Cycle 1
  To determine the pharmacokinetics of oral aza-TdC
To document preliminary evidence of aza-TdCyd activity | Cycle 1 and 2
  To document preliminary evidence of aza-TdC activity
To determine effect of study treatment on re-expression of select genes silenced by methylation in circulating tumor cells | Cycle 1 and 2
  To determine effect of study treatment on re-expression of select genes silenced by methylation in circulating tumor cells
To determine the effects of Aza-TdC on DNA damage response (DDR) signaling and on genome-wide DNA methylation in tumor biopsy tissue | Pre-treatment, Cycle 1 Day 2, Cycle 2 Day 10
  To determine the effects of Aza-TdC on DNA damage response (DDR) signaling and on genome-wide DNA methylation in tumor biopsy tissue

CONTACTS AND LOCATIONS:
Overall Officials: James H Doroshow, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Background] Cowan LA, Talwar S, Yang AS. Will DNA methylation inhibitors work in solid tumors? A review of the clinical experience with azacitidine and decitabine in solid tumors. Epigenomics. 2010 Feb;2(1):71-86. doi: 10.2217/epi.09.44. PMID 22122748
- [Background] Thottassery JV, Sambandam V, Allan PW, Maddry JA, Maxuitenko YY, Tiwari K, Hollingshead M, Parker WB. Novel DNA methyltransferase-1 (DNMT1) depleting anticancer nucleosides, 4'-thio-2'-deoxycytidine and 5-aza-4'-thio-2'-deoxycytidine. Cancer Chemother Pharmacol. 2014 Aug;74(2):291-302. doi: 10.1007/s00280-014-2503-z. Epub 2014 Jun 8. PMID 24908436
- [Background] Tiwari KN, Cappellacci L, Montgomery JA, Secrist JA 3rd. Synthesis and anti-cancer activity of some novel 5-azacytosine nucleosides. Nucleosides Nucleotides Nucleic Acids. 2003 Dec;22(12):2161-70. doi: 10.1081/ncn-120026872. PMID 14714764
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2018-C-0014.html